CLINICAL TRIAL: NCT00006098
Title: A Phase I Study of PS-341 in Patients With Hematologic Malignancies
Brief Title: PS-341 in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-031; CDR0000068105 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1827
Record Dates: First submitted 2000-08-03; First posted 2004-03-17 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent adult Hodgkin lymphoma; refractory multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; previously treated myelodysplastic syndromes; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory, with Excess of Blasts; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: PS-341 may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase I trial to study the effectiveness of PS-341 in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose-limiting toxicity of PS-341 in patients with hematologic malignancies. II. Determine the pharmacodynamics of this drug in these patients. III. Determine response to this drug in these patients. IV. Determine the correlation between response of malignancies and proteasome inhibition and apoptosis in peripheral blood mononuclear cells (PBMC) of these patients. V. Determine the correlation between therapy toxicity and proteasome inhibition and apoptosis in PBMC of these patients. VI. Determine the effect of this drug on other molecular markers (i.e., BCL-2 in follicular lymphoma patients and t9;22/BCR/ABL in chronic lymphocytic leukemia patients). VII. Determine the correlation between interleukin-6 serum levels in multiple myeloma patients and drug dosing, toxicity of therapy, extent of protease inhibition, response to therapy, and apoptosis in PBMC of these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients receive PS-341 IV over 30 minutes on days 1, 4, 8, 11, 15, 18, 22, and 25 followed by a 2-week rest. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of PS-341 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed hematologic malignancy including: Acute myeloid leukemia Chronic myelogenous leukemia Acute lymphoblastic leukemia Chronic lymphocytic leukemia Hodgkin's disease Non-Hodgkin's lymphoma Multiple myeloma Myelodysplastic syndrome subtypes: Refractory anemia with excess blasts (RAEB) RAEB in transformation Refractory to standard treatment or no curative therapy available Measurable disease Not eligible for higher priority study

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 6 weeks Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,000/mm3 Platelet count at least 50,000/mm3 Hematocrit at least 25% Hepatic: SGOT and SGPT less than 2.5 times upper limit of normal (ULN) Bilirubin less than 1.5 times ULN Renal: Creatinine clearance greater than 50 mL/min Cardiovascular: No acute ischemia or new conduction system abnormalities by EKG No prior myocardial infarction within past 6 months No New York Heart Association class III or IV congestive heart failure Other: Febrile episodes up to 38.5 degrees C due to tumor fever allowed No concurrent active infection No grade 1 or greater National Cancer Institute common toxicity criteria No serious medical or psychiatric condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy No concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: At least 2 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Soignet, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States